CLINICAL TRIAL: NCT03315663
Title: Effectiveness and Safety of a Smartphone-Assisted Personalized Intervention Program to Reduce Diabetes Risk in Adults With Prediabetes: a Multi-Center, Open-Label Randomized Controlled Trial - Main Study
Brief Title: Personalized Smartphone-assisted Coaching System to Improve Glucose Homeostasis in Adults With Prediabetes - Main Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn due to budgetary and other constraints.
Sponsor: Johns Hopkins University (Other)
Collaborators: Sweetch Health, Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00099813
Record Dates: First submitted 2017-09-05; First posted 2017-10-20 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Prediabetes; Hyperglycemia; Postprandial Hyperglycemia; Impaired Glucose Tolerance; Impaired Fasting Glucose
Keywords: Mobile Health
MeSH Terms: conditions — Prediabetic State; Hyperglycemia; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: This Pivotal Study will be a multicenter, parallel group, open-label randomized controlled trial with a planned period of 12-month follow-up with the primary effectiveness endpoint assessed at 6 months to compare Sweetch's mHealth Personalized Intervention Program (PIP) to usual care for adults with prediabetes. We intend to enroll 155 subjects in each arm, for a total of 310 subjects in this Study. Subjects will attend a total of 3 visits during the study period with point-of-care measurement of A1C at each study visit (0, 6, and 12 months). A difference in change in A1c of 0.1 between the intervention and control arms and in favor of the intervention arm will be considered clinically meaningful.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sweetch App + DBWS (Active Comparator): Participants receive usual care for prediabetes management. In addition, participants will be randomized to receive the Sweetch app plus weight monitoring via digital body weight scale (DBWS).
  Interventions: Other: Sweetch App & DBWS
- Sweetch App Alone (Active Comparator): Participants receive usual care for prediabetes management. In addition, participants will be randomized to receive the Sweetch app alone.
  Interventions: Other: Sweetch App Alone

INTERVENTIONS:
Other: Sweetch App & DBWS — Usual care for prediabetes management, Sweetch app, weight monitoring via digital body weight scale (DBWS).
  Arms: Sweetch App + DBWS
Other: Sweetch App Alone — Usual care for prediabetes management, Sweetch app alone.
  Arms: Sweetch App Alone

SUMMARY:
Sweetch is a personalized mobile-health platform coaching system (mobile phone app) designed to promote adherence to physical activity guidelines for people with prediabetes.

DETAILED DESCRIPTION:
The mobile phone app Sweetch seeks to increase leisure time physical activity rather than formal exercise through the use of a behavioral analytics engine that continuously process various aspects of the user's life habits, taking into account the user's demographics, behavioral change status, schedule, actual activity patterns, and more. The rationale behind this approach is that long-term adherence and patient engagement are more likely to be achieved when demands on manual user data entry are kept at a minimum. Compared to similar smartphone-assisted prevention apps, there are two novel features of the Sweetch app that may increase its efficacy. First, it uses a "just-in-time" adaptive intervention" approach that tailors recommendations to the user's day-to-day routine and his or her readiness for behavioral change. Second, and most importantly, it requires no direct involvement by the user, since all the necessary data is collected using built-in tracking pedometers, accelerometer and Global Positioning System (GPS) sensors on smartphones. In contrast, interventions that focus on dietary changes (i.e. calorie reduction, change in macronutrient content), require active user tracking at every meal, which is difficult to maintain in the long-term even with the use of sophisticated, electronic calorie counting tools. For these reasons, the Sweetch app may achieve greater long-term adherence, which is usually a limiting factor to efficacy of mobile health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 -75 years with prediabetes (fasting Blood Glucose (BG) 100-125 mg/dl, A1C 5.7% - 6.4%, or 2 hour BG of 140-199 mg/dl following 75-gram oral glucose tolerance test)
* Body mass index 24 - 40 kg/m2
* English speaker
* Smartphone user (Android or Apple 5s and above)

Exclusion Criteria:

* Currently doing more than 150 minutes/week of moderate/vigorous physical activity
* Presence of medical conditions that prevent adoption of moderate physical activity
* Use of any glucose-lowering or weight loss medications within the previous 3 months
* Current pregnancy (self-reported) or planning pregnancy during study period (self-reported)
* Presence of any condition that can result in spurious A1C readings (e.g. anemia [hemoglobin level below lower limit of normal] secondary to iron, vitamin B12, or folate deficiencies; hemoglobinopathies)
* Use of systemic glucocorticoids
* Use of antipsychotic medications (stable doses for at least three months of anti-depressants or anti-anxiety drugs will be allowed)
* Severe mental illness or learning disability
* Current participation in another clinical trial
* Liver enzymes >3 x upper limit of normal
* Poor literacy (REALM-R score of 6 or less)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Safety of Sweetch's PIP compared to usual care to lower A1C | 2 years
  Administration of study intervention will be halted when 3 grade 3 Adverse Events (AEs) determined to be "probably related" are reported to the Data Coordinating Center (DCC). The DCC will notify study sponsor & investigators immediately when the third grade 3 event is reported & enrollment screens will stop accepting new study participants. Study sponsor will inform the Data Safety and Monitoring Board (DSMB) members within 24 hours of this occurrence & will provide DSMB with AE listing reports. The DSMB will convene an ad hoc meeting by teleconference or in writing as soon as possible. The DSMB will provide recommendations for proceeding with the study to study sponsor. If Sweetch Health determines that an unanticipated adverse device effect presents an unreasonable risk to subjects, investigations or parts of investigations presenting that risk will be terminated as soon as possible.
Effectiveness of Sweetch's PIP compared to usual care to lower A1C | 2 years
  A1C is a continuous measure expressed in units of % and mmol/mol. Change in A1C will be calculated by subtracting the 6-month result from the baseline result. The primary effectiveness endpoint will be analyzed using linear regression models, where change in A1C at 6 months will be the dependent variable and treatment group will be the primary predictor variable. The baseline value of the outcome measure will be included as a covariate.

SECONDARY OUTCOMES:
Evaluation of whether intervention increases physical activity. | 12 months
  Through the use of built-in accelerometers and pedometers on smartphones, the study will evaluate the percentage of weekly activity goals (individualized per subject) achieved per subject (range from 60 minutes to 150 minutes per week), proportion of subjects achieving 150 minutes of weekly activity taken as the average of months 4-6 at the 6-month time point, and average of months 7-12 at the 12-month time point. In addition, mean minutes of physical activity per week will be evaluated over intervals between study time points. Physical activity measures will be reported only in the intervention arm, since tracking of physical activity will not be possible in the control arm.
Evaluation of whether intervention reduces weight. | 12 months
  Users update manually or weight data is synced from the digital scale. Data points measured are net weight change from baseline to 6 and 12 months; percentage weight change from baseline to 6 and 12 months; and proportion of subjects achieving 5% body weight loss at 6 and 12 months.
Evaluation of whether intervention reduces waist circumference. | 12 months
  Waist circumference will be measured using a flexible tape measure according to the technique recommended by the American Society for Nutrition. We will evaluate percentage change in waist circumference from baseline to 6 and 12 month time points. The null hypothesis is that there is no difference between percentage change at 6 and 12 months between the intervention and control groups and the alternative hypothesis is that there is a greater percentage change in waist circumference from baseline in the intervention group.
Evaluation of whether intervention reduces blood pressure. | 12 months
  Blood pressure will be measured in accordance with recommendations by the American Heart Association. Changes in systolic and diastolic blood pressure from baseline to 6 and 12 months. Systolic (SBP) and diastolic blood pressure (DBP) will be evaluated as separate continuous measures. The null hypothesis is that changes in SBP and DBP are no different between groups at both time points and the alternative hypothesis is that there is a greater reduction in SBP and DBP in the intervention group. Assuming a variance of 10.1 for change in SBP38 and a change of -1 mmHg in the control arm, the study would have 83% power to detect a between-group difference of 4 mmHg in SBP, which would be considered clinically meaningful. Assuming a variance of 7 for change in DBP and a change of -1 mmHg in the control arm38, the study would have 81% power to detect a between-group difference of 2.7 mmHg in DBP, which would be considered clinically meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S. Dobs, MD MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Reading Health System, Reading, Pennsylvania

IPD SHARING:
Plan to Share IPD: No